CLINICAL TRIAL: NCT05266443
Title: The Efficacy of Lactobacillus-containing Cultured Milk Drink in Alleviating Subthreshold Depression Among Adults With Irritable Bowel Syndrome
Brief Title: Lactobacillus-containing Cultured Milk Drink Alleviates Depression Score Among Adults With Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Cotra Enterprises Sdn. Bhd. (Unknown)
Responsible Party: Principal Investigator, PROF DR RAJA AFFENDI RAJA ALI, Consultant Physician & Gastroenterologist, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UKM PPI/111/8/JEP-2019-312
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Irritable Bowel Syndrome With Subthreshold Depression
Keywords: irritable bowel syndrome; subthreshold depression; probiotics; IBS; subclinical depression
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomized and parallel study involving patients with IBS who attended gastroenterology clinics at Universiti Kebangsaan Malaysia Medical Center (UKMMC). The recruited subjects will be categorized according to their CESD-R scores and randomly allocated into receiving either placebo or probiotic-containing cultured milk drink for 12 weeks.
Who Masked: Participant, Investigator
Masking Description: Both investigators and subjects will be blinded to the treatment products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Irritable bowel syndrome with normal mood receiving placebo (Placebo Comparator): A total of 35 patients diagnosed with IBS as per Rome IV criteria who scored CESD-R less than 16 will be supplemented with placebo drinks.
  Interventions: Dietary Supplement: Placebo cultured milk drink
- Irritable bowel syndrome with normal mood receiving probiotics (Active Comparator): A total of 35 patients diagnosed with IBS as per Rome IV criteria who scored CESD-R less than 16 will be given lactobacillus-containing cultured milk drinks.
  Interventions: Dietary Supplement: Lactobacillus containing cultured milk drink
- Irritable bowel syndrome with subthreshold depression receiving placebo (Placebo Comparator): A total of 35 patients diagnosed with IBS as per Rome IV criteria who scored CESD-R of 16 or above will be supplemented with placebo drinks.
  Interventions: Dietary Supplement: Placebo cultured milk drink
- Irritable bowel syndrome with subthreshold depression receiving probiotics (Experimental): A total of 35 patients diagnosed with IBS as per Rome IV criteria who scored CESD-R of 16 or above will be given lactobacillus-containing cultured milk drinks.
  Interventions: Dietary Supplement: Lactobacillus containing cultured milk drink

INTERVENTIONS:
Dietary Supplement: Lactobacillus containing cultured milk drink — Each bottle of 125ml cultured milk drink contains a billion colony forming unit (CFU) Lactobacillus acidophillus (LA-5) and Lactobacillus paracasei (L. CASEI-01). Each patient will be given 2 bottles to consume daily for a period of 12 weeks.
  Arms: Irritable bowel syndrome with normal mood receiving probiotics; Irritable bowel syndrome with subthreshold depression receiving probiotics
Dietary Supplement: Placebo cultured milk drink — The placebo prepared was identical to the probiotic-containing product in terms of color, taste and packaging. However, there is no trace of live microorganism in this product.
  Arms: Irritable bowel syndrome with normal mood receiving placebo; Irritable bowel syndrome with subthreshold depression receiving placebo

SUMMARY:
Irritable bowel syndrome (IBS) is frequently associated with any form of psychiatric comorbidities including subthreshold or subclinical depression. Modification of gut ecology with probiotics has implicitly improved IBS and depressive symptoms. However, the efficacy of probiotics on IBS with existing subthreshold depression remain elusive. Therefore, the aim of this study is to evaluate the effects of lactobacillus-containing cultured milk drink on depression scores in adults diagnosed with IBS.

DETAILED DESCRIPTION:
A total of 140 subjects who fulfilled Rome IV criteria for IBS will be recruited from a tertiary medical centre and among public volunteers. The depression status and categories will be assessed using the Centre Epidemiologic Studies Depression Scale Revised questionnaire (CESD-R): normal mood (score<16), or subthreshold depression (score>16). The subjects are randomised and blinded into four groups: Group A (Normal mood with placebo, n=35), Group B (Normal mood with probiotics, n=35), Group C (Subthreshold depression with placebo, n=35) and Group D (Subthreshold depression with probiotics, n=35). The subjects will be instructed to consume two bottles of cultured milk drink daily for 12 weeks. The probiotic cultured milk drinks contained 10^9 cfu L. CASEI-01 and LA-5. The severity of depression will be measured using Patient Health Questionnaire (PHQ-9) at pre- and post-12-week intervention. Secondary outcome on IBS symptoms severity will be assessed with IBS Symptoms Severity Score (IBS-SSS) and IBS Quality of Life (IBS-QOL).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years old,
* Meet ROME IV criteria for irritable bowel syndrome,
* Consented to participate in the study.

Exclusion Criteria:

* Lactose intolerance,
* Gastrointestinal disorders such as inflammatory bowel diseases, liver diseases, pancreatic diseases or malignancies,
* Any neurological diseases or malignancies,
* Pregnant and lactating mothers,
* Any metabolic diseases such as hypertension, hypercholesterolaemia, diabetes mellitus, hyper- and hypothyroidism.
* Known psychiatric diagnoses or/and consume psychotropic drugs,
* Ongoing electroconvulsive therapy (ECT),
* Consumption of antibiotics, probiotics, prebiotics, symbiotics products, laxatives, antispasmodics, and/or anticholinergics who refuse to consent for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Depression score | 12 weeks
  The Centre for Epidemiologic Studies Depression Scale Revised Version (CESD-R) will be used to classify the patients according to their depression status.
Depression severity scale | 12 weeks
  The Patient Health Questionnaire-9 (PHQ-9) will be used to assess the severity scale for the patients.

SECONDARY OUTCOMES:
Quality of life score | 12 weeks
  The life quality of patients will be measured using the Irritable bowel syndrome Quality of Life Questionnaire (IBS-QOL).
IBS severity score | 12 weeks
  Any changes in gastrointestinal symptoms severity related to IBS will be quantify using the Irritable bowel syndrome Severity Scoring System (IBS-SSS).
Acute stress biomarker | 12 weeks
  Morning blood sample will be collected to measure serum cortisol level among patients with IBS.
Depression biomarker | 12 weeks
  Blood samples collected will be analysed to measure the serum serotonin level of patients with IBS.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Raja Affendi Raja Ali, Principal Investigator — Gastroenterology Unit, Faculty of Medicine, Universiti Kebangsaan Malaysia, Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia, Bandar Tun Razak, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No